CLINICAL TRIAL: NCT06732323
Title: A Randomized, Open-label, Phase III Study of ESG401 Versus Investigator's Choice Chemotherapy as First-line Treatment in Patients With Unresectable Recurrent or Metastatic Triple-Negative Breast Cancer
Brief Title: A Phase III Study of ESG401 for Unresectable Recurrent or Metastatic Triple-Negative Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESG401-302
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2024-12

CONDITIONS: Triple-Negative Breast Cancer (TNBC)
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESG401 for injection (Experimental): IV infusion on day 1, 8 and15 of each 28 day cycle
  Interventions: Drug: ESG401
- Investigator's Choice Chemotherapy (Active Comparator): If no prior taxane, or prior taxane in the (neo)adjuvant setting and disease-free interval (DFI) >12 months: paclitaxel or nab-paclitaxel. Note: If subjects are intolerant or contraindicated to receive paclitaxel or albumin-paclitaxel, the investigator may choose other chemotherapy options listed in the study protocol) If prior taxane and DFI ≤ 12 months: capecitabine, eribulin. If known BRCA1/2 mutation: carboplatin
  Interventions: Drug: Investigator's Choice Chemotherapy

INTERVENTIONS:
Drug: ESG401 — IV infusion on day 1,8, and 15 of each 28 day cycle
  Arms: ESG401 for injection
Drug: Investigator's Choice Chemotherapy — Paclitaxel, Nab-paclitaxel, Capecitabine, Eribulin, or Carboplatin
  Arms: Investigator's Choice Chemotherapy

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of ESG401 as first-line treatment in patients with unresectable recurrent or metastatic triple-negative breast cancer.

DETAILED DESCRIPTION:
This is a randomized, open-label, multicenter Phase 3 study to evaluate ESG401 versus Investigator's Choice Chemotherapy (ICC) as first-line treatment in subjects with unresectable recurrent or metastatic triple-negative breast cancer.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males or females aged ≥ 18 years ;
2. Histologically and/or cytologically confirmed TNBC;
3. De novo metastatic or relapsed ≥ 6 months post completion of treatment with curative intent;
4. No prior systemic anti-cancer therapy for unresectable recurrent or metastatic disease;
5. Participants whose tumours are PD-L1-negative, or Participants whose tumours are PD-L1-positive and have relapsed after prior PD-1/PD-L1 inhibitor therapy for early-stage breast cancer, or comorbidities precluding PD-1/PD-L1 inhibitor therapy;
6. Eligible for the chemotherapy options listed as investigator's choice chemotherapy (paclitaxel, nab-paclitaxel, capecitabine, eribulin, or carboplatin) as assessed by the investigator;
7. At least one measurable lesion per RECIST v1.1;
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 with no worsening within 2 weeks prior to randomization;
9. A life expectancy of at least 12 weeks;
10. Adequate organ and bone marrow function.

Key Exclusion Criteria:

1. Use of any investigational anti-cancer drug within 28 days or 5 half-lives before the first investigational product administration.
2. Toxicities from prior anti-tumor therapy not recovering to ≤ Grade 1.
3. Prior topoisomerase I inhibitor therapy, including antibody-drug conjugate(ADC) therapy, or prior TROP2 targeted therapy.
4. New thromboembolic events, intestinal obstruction, gastrointestinal bleeding or perforation within 6 months.
5. Subjects with symptomatic or untreated CNS metastases, or those requiring ongoing treatment for CNS metastases.
6. Patients with Primary CNS malignancy, or patients with other malignancies within 3 years prior to the first dose.
7. Patients with uncontrollable systemic diseases.
8. Patients with gastrointestinal diseases (such as chronic gastritis, chronic enteritis or gastric ulcers), or with a previous history of severe or chronic diarrhea.
9. Subjects with clinically significant cardiovascular disease.
10. Human Immunodeficiency Virus (HIV) infection.
11. Active hepatitis B or hepatitis C.
12. Known immediate or delayed hypersensitivity reaction to irinotecan or other camptocampin derivatives such as topotecan or to have had grade≥3 gastrointestinal reactions associated with irinotecan, or allergies, or to any investigational drug or excipient ingredient.
13. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) assessed by Blinded Independent Central Review (BICR) | Randomization up to approximately 28 months
  Defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on BICR or death due to any cause, whichever occurs first.
Overall Survival (OS) | Randomization up to approximately 41 months
  Defined as the time from randomization until the date of death due to any cause.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) assessed by Investigator | Randomization up to approximately 28 months
  Defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on investigator or death due to any cause, whichever occurs first.
Objective Response Rate (ORR) assessed by Blinded Independent Central Review (BICR) | Randomization up to approximately 28 months
  Defined as the percentage of patients who achieve complete response(CR) or partial response (PR), as assessed by BICR per RECIST 1.1
Disease control rate (DCR) assessed by Blinded Independent Central Review (BICR) | Randomization up to approximately 28 months
  Defined as the percentage of patients who achieve CR, PR or stable disease (SD), as assessed by BICR per RECIST 1.1
Duration of Response (DoR) assessed by Blinded Independent Central Review (BICR) | Randomization up to approximately 28 months
  Defined as the time from the date of first documented CR or PR until date of documented disease progression per RECIST 1.1, as assessed by BICR or death due to any cause, whichever occurs first.
Time to Response (TTR) assessed by Blinded Independent Central Review (BICR) | Randomization up to approximately 28 months
  Defined as the time from the date of randomization until the first documentation of CR or PR as assessed by BICR per RECIST 1.1.
Objective Response Rate (ORR) assessed by Investigator | Randomization up to approximately 28 months
  Defined as the percentage of patients who achieve complete response(CR) or partial response (PR), as assessed by investigator per RECIST 1.1
Disease control rate (DCR) assessed by Investigator | Randomization up to approximately 28 months
  Defined as the percentage of patients who achieve CR, PR or stable disease (SD), as assessed by investigator per RECIST 1.1
Duration of Response (DoR) assessed by Investigator | Randomization up to approximately 28 months
  Defined as the time from the date of first documented CR or PR until date of documented disease progression per RECIST 1.1, as assessed by investigator or death due to any cause, whichever occurs first.
Time to Response (TTR) assessed by Investigator | Randomization up to approximately 28 months
  Defined as the time from the date of randomization until the first documentation of CR or PR as assessed by investigator per RECIST 1.1.
Quality of life evaluated using the NCC-BC-A scale | Randomization up to approximately 28 months
  To assess the impact of ESG401 on disease related symptoms and quality of life of patients using the NCC-BC-A scale
Adverse events(AEs) and severe adverse events (SAEs) | From signing the ICF up to last dose plus 30 days
  Incidence and severity of AEs and SAEs (per CTCAE 5.0), and clinically significant abnormal laboratory findings
Clearance | Randomization up to approximately 28 months
  Mean population clearance will be derived from pooled data of drug concentrations. Covariates of influence on drug clearance will be incorporated within a population pharmacokinetic model.
Volume of distribution | Randomization up to approximately 28 months
  Mean population volume of distribution will be derived from pooled data of drug concentrations. Covariates of influence on volume of distribution will be incorporated within a population pharmacokinetic model.
Anti-drug Antibodies | Randomization up to approximately 28 months
  Incidence of anti-drug antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Ma, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No